CLINICAL TRIAL: NCT04910711
Title: Contraceptives and Dolutegravir-based ART
Brief Title: Investigating the Interaction Between Two Long-acting Reversible Methods of Contraception and Dolutegravir, a Treatment for HIV
Acronym: CODA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Botswana Harvard AIDS Institute Partnership (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Chelsea Morroni, Principal Investigator, Botswana Harvard AIDS Institute Partnership
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UBR/RES/IRB//BIO/236
Record Dates: First submitted 2021-05-24; First posted 2021-06-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Human Immunodeficiency Virus; Contraception; ART
Keywords: Contraception; HIV; Antiretroviral Therapy; Dolutegravir; Drug interactions; Etonogestrel implant; Contraceptive implant; DMPA injection; Contraceptive injection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Levonorgestrel; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- DTG/LNG (Active Comparator): Receiving dolutegravir-based antiretroviral therapy and initiating the levonorgestrel implant
  Interventions: Drug: Dolutegravir; Drug: Levonorgestrel implant
- NEG/LNG (Other): HIV negative, not receiving antiretroviral therapy and initiating the levonorgestrel implant
  Interventions: Drug: Levonorgestrel implant
- DTG/MPA (Active Comparator): Receiving dolutegravir-based antiretroviral therapy and the depot medroxyprogesterone acetate injection
  Interventions: Drug: Dolutegravir; Drug: Depo medroxyprogesterone acetate injection
- NEG/MPA (Other): HIV negative, not receiving antiretroviral therapy and receiving the depot medroxyprogesterone acetate injection
  Interventions: Drug: Depo medroxyprogesterone acetate injection

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir-based antiretroviral therapy
  Arms: DTG/LNG; DTG/MPA
Drug: Levonorgestrel implant — Women initiating the levonorgestrel implant
  Arms: DTG/LNG; NEG/LNG
Drug: Depo medroxyprogesterone acetate injection — Women initiating the depo medroxyprogesterone acetate injection
  Arms: DTG/MPA; NEG/MPA

SUMMARY:
It is important to make sure that women have access to effective methods of contraception to prevent pregnancy so that they can make choices about when and if they will have their first or next child. Some of the most effective methods of contraception are the long-acting, reversible methods of contraception (LARCS), including the contraceptive implant and the contraceptive injection. In areas of the world where there are high numbers of people living with HIV, providing contraception to women is sometimes complicated, as there are known to be interactions between some of the medications that treat HIV and some hormonal methods of contraception. One medication to treat HIV, dolutegravir, is now one of the first-line treatments for HIV in Botswana, and more and more women of childbearing age are taking dolutegravir to treat HIV. At the moment, there is limited information on whether or not there are interactions between dolutegravir (the HIV medication) and the contraceptive implant or the contraceptive injection, two commonly used methods of contraception in Botswana. The main purpose of this study is to find out if women using contraception and also taking dolutegravir have lower levels of contraceptive hormone in their blood compared to women taking no HIV treatment. The study hypothesis is that there is no interaction between dolutegravir and the contraceptive implant or injection.

In this study, levels of hormone from the injection or the implant will be measured in women living with HIV who take dolutegravir and compared to hormone levels in women who do not have HIV and who have never taken any medications to treat HIV. Women will be counselled about all of the possible methods of contraception (including the pill, the injection, the implant and the copper intrauterine device (or coil/loop)) that are available and will be empowered to make their own decision about the method of contraception they feel will be best for them. Women who choose the implant or the injection will be invited to enrol in the study; and will be categorised into one of four groups, based on whether or not they are living with HIV and taking dolutegravir. At several time points, women will have blood tests to check the level of hormone from the implant or the injection, over a course of 12 weeks for women starting the injection and 24 weeks for women starting the implant. Women will also be asked to complete a short questionnaire about any side effects from the contraception including changes to bleeding patterns. At the end of the 12 weeks (for women starting the injection) or 24 weeks (for women starting the implant), the results from these blood samples will be analysed to see how the levels of the hormone in their blood changed over time. The study will also look at whether the levels of dolutegravir (the HIV medication) changed over time. These results will be compared between women living with HIV taking dolutegravir and women without HIV who have never taken dolutegravir to see whether there is any interaction between dolutegravir and the hormonal contraceptive implant or contraceptive injection.

DETAILED DESCRIPTION:
This study will evaluate whether dolutegravir (DTG)-based antiretroviral therapy (ART) given with two widely used hormonal contraceptives avoid pharmacokinetic drug-drug interactions that lead to reduced levels of hormonal concentrations and could, thus, reduce contraceptive effectiveness. Two highly effective and commonly used methods of hormonal contraception in African settings will be studied: the levonorgestrel (LNG) sub-dermal contraceptive implant and the depot medroxyprogesterone acetate (DMPA) injectable contraceptive.

Overall, the investigators hypothesise that the plasma concentrations of the studied hormonal contraceptives in women living with HIV-1 and taking DTG-based ART will be equivalent to concentrations in HIV-negative, ART naïve women.

Specific Aims:

Specific Aim 1: To compare plasma LNG concentrations among (a) levonorgestrel contraceptive implant-users in Botswana receiving DTG-based ART and (b) HIV-negative, ART naïve levonorgestrel contraceptive implant users.

Specific Aim 2: To compare plasma medroxyprogesterone acetate (MPA) concentrations among (a) DMPA injectable-users in Botswana receiving DTG-based ART and (b) HIV-negative, ART naïve DMPA injectable users.

Specific Aim 3: To compare the trough plasma concentrations of DTG before and after contraceptive use to understand how LNG and DMPA may affect DTG exposure.

Specific Aim 4: To determine if the LNG implant and DMPA injectable inhibit ovulation in the presence of DTG.

Specific Aim 5: To evaluate safety, tolerability, bleeding patterns and contraceptive method continuation with concomitant LNG implant or DMPA injectable, compared to controls (HIV negative, ART naïve women).

ELIGIBILITY:
Inclusion Criteria:

* Sex female
* Age 18-45 years
* Desire to use LNG implant (for at least 6 months) or for at least one cycle of use of DMPA injectable (3 months), following comprehensive client-centered contraceptive counselling
* Willing and able to initiate the LNG implant or the DMPA injectable at enrolment visit or soon thereafter
* Participants who are engaging in sexual activity that could lead to pregnancy must agree to use a non-hormonal method of contraception, in addition to the LNG implant or DMPA injectable, while participating in the study. Acceptable contraceptives include: condoms (male or female); diaphragm or cervical cap with spermicide; non-hormonal intrauterine device; bilateral tubal ligation; and male partner vasectomy
* No acute infections or other opportunistic diseases requiring systemic medication of hospitalisation within 14 days prior to study entry
* The following laboratory values:

  * Haemoglobin ≥8.0 g/dL
  * Creatinine clearance >60 mL/min/1.73m2
  * Aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) <2.5 x upper limit of normal ULN
  * Alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) <2.5 x ULN
  * Platelet count ≥50,000 platelets/mm3
* Last menstrual period ≤35 days prior to study entry
* No sexual activity that could lead to pregnancy since last menstrual period without contraception (condoms, male or female); diaphragm or cervical cap with spermicide; non-hormonal intrauterine device; bilateral tubal ligation; and male partner vasectomy), as reported by study participant and assessed by study clinician
* Negative serum or urine pregnancy test at screening and study enrolment
* Willing to undergo questionnaires, examinations and phlebotomy per schedule for the duration of the study period
* Able to consent for study participation in English or Setswana

For HIV-positive participants:

* Documented HIV-1 infection
* Using DTG-based ART (DTG 50mg once daily co-administered with 2 NRTIs (emtricitabine/tenofovir or lamivudine/tenofovir)
* DTG-based ART use (for at least 30 days prior to contraceptive method initiation). On stable regimen containing DTG and 2 NRTIs for ≥ 30 days without gaps in adherence in the last 30 days prior to study entry, and no known plans to change ART regimen for the duration of the study
* Most recent HIV plasma RNA below lower limit of quantitation of the assay used per standard of care

Exclusion Criteria:

* Sex male
* Women <18 years
* Any contraindication (WHO Medical Eligibility Criteria for Contraceptive Use Category 3 or 4) to receiving the selected contraceptive method, based on WHO Medical Eligibility Criteria for Contraceptive Use (24)
* Postpartum less than 6 weeks
* Currently breastfeeding
* Currently pregnant or intends to become pregnant during the study
* The following laboratory values:

  * Hemoglobin <8.0 g/dL
  * Creatinine clearance ≤60 mL/min/1.73m2
  * Aspartate transaminase (AST; SGOT) ≥2.5 x ULN
  * Alanine transaminase (ALT; SGPT) ≥2.5 x ULN
  * Platelet count <50,000 platelets/mm3
* Receipt of DMPA during the 120 days or norethisterone enanthate (NET-EN) during the 60 days prior to study entry
* Initiated the LNG implant prior to study entry
* Receipt of other hormonal treatments (e.g., oral contraceptives, contraceptive vaginal ring, contraceptive patch, or oral hormone replacement therapy) within the 30 days prior to study entry
* The study puts the participant at unacceptable risk based on the judgment of the study staff
* Known allergy/sensitivity or any hypersensitivity to components of study medication(s) or their formulation
* Active drug or alcohol use or dependence that would interfere with adherence to study requirements
* Concomitant use of drugs known to be contraindicated with LNG or MPA
* Use of any drugs known to: 1) induce CYP3A4 system within 30 days or 2) inhibit the CYP3A4 system with one week prior to enrolment visit
* Use or anticipated use of concomitant enzyme-inducing drugs, including but not limited to rifampicin for tuberculosis treatment and anti-convulsant medications (e.g., phenytoin, carbamazepine, barbiturates, primidone, topiramate, oxcarbazepine, felbamate)
* Unwilling to attend study visits or adhere to study visit procedures
* Unable to consent

For HIV-positive participants:

* Self-reported non-adherence to ART
* Concomitant use of drugs known to be contraindicated with DTG or medicinal products that reduce DTG exposure (e.g. magnesium/ aluminium-containing antacid, iron and calcium supplements, multivitamins and inducing agents, rifampicin, St. John's wort and anti-epileptic medicinal products carbamazepine, oxcarbazepine, phenytoin and phenobarbital)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
24-week levonorgestrel area under the concentration-time curve (AUC) | The AUC0-24 weeks will be calculated at 24 weeks from participant enrolment, using levonorgestrel concentrations measured at 0, 2, 4, 8, 12, 16 and 24 weeks post-levonorgestrel implant initiation.
  The AUC of levonorgestrel over 0-24 weeks will be estimated in women initiating the levonorgestrel implant. The levonorgestrel AUC0-24 weeks will be compared between women living with HIV receiving dolutegravir-based antiretroviral therapy and HIV-negative women who have never taken antiretroviral therapy.
12-week medroxyprogesterone acetate AUC | The AUC0-12 weeks will be calculated at 12 weeks from participant enrolment, using medroxyprogesterone acetate concentrations measured at 0, 2, 4, 8, 10 and 12 weeks post-DMPA injection initiation.
  The AUC of medroxyprogesterone acetate over 0-12 weeks will be estimated in women initiating the depot medroxyprogesterone acetate injection. The medroxyprogesterone acetate AUC0-12 weeks will be compared between women living with HIV receiving dolutegravir-based antiretroviral therapy and HIV-negative women who have never taken antiretroviral therapy.

SECONDARY OUTCOMES:
Cmin for levonorgestrel, medroxyprogesterone acetate and dolutegravir | 24 weeks (LNG) or 12 weeks (MPA)
  Minimum plasma drug concentration (Cmin)
Cmax for levonorgestrel, medroxyprogesterone acetate and dolutegravir | 24 weeks (LNG) or 12 weeks (MPA)
  Maximum plasma drug concentration (Cmax)
CL/F of levonorgestrel, medroxyprogesterone acetate and dolutegravir | 24 weeks (LNG) or 12 weeks (MPA)
  Apparent oral clearance (CL/F)
Ovulation | 24 weeks (LNG) or 12 weeks (MPA)
  Number of participants with endogenous progesterone concentrations above the threshold for ovulation at all time points up to week 24 (LNG) or week 12 (MPA)
Safety, tolerability, side effects and bleeding patterns | 24 weeks (LNG) or 12 weeks (MPA)
  Number of participants with reported adverse events or side effects (e.g. changes to bleeding pattern) over the course of the study.
Contraception method continuation | 24 weeks (LNG) or 12 weeks (MPA)
  Number of participants who chose to continue method of contraception at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Morroni, PhD MBChB, Principal Investigator — Botswana Harvard AIDS Institute Partnership
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No